CLINICAL TRIAL: NCT03792971
Title: Phase 1, Open-label, One-arm, Fixed-sequence Study to Evaluate the Effects of 90 mg Intravenous Infusions of GC4419 on the Single Dose Pharmacokinetics of Dextromethorphan in Healthy Adult Subjects
Brief Title: Study to Evaluate the Effects of 90 mg Intravenous Infusions of GC4419 on the Single Dose Pharmacokinetics of Dextromethorphan in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI-4419-005
Record Dates: First submitted 2018-12-21; First posted 2019-01-04 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dextromethorphan; avasopasem manganese

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fixed Sequence (Experimental)
  Interventions: Drug: Dextromethorphan HBr; Drug: GC4419

INTERVENTIONS:
Drug: Dextromethorphan HBr — A single 60 mg dose of DM capsules liquid-filled on Day 1 and Day 3
Drug: GC4419 — Daily 90 mg IV infusions over 60 minutes on Day 3 and Day 4

SUMMARY:
This will be a single center, phase 1, open-label, fixed-sequence study under fasting conditions to evaluate the effect of 90 mg intravenous (IV) infusions of GC4419 on the single-dose pharmacokinetic (PK) of dextromethorphan (DM) capsules liquid filled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker, ≥ 18 and ≤ 55 years of age, with BMI > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Females of childbearing potential must be willing to use acceptable contraceptive method throughout the study and for 30 days after the last study drug administration:
4. Male subjects must be willing to use acceptable contraceptive method from the first dosing until at least 90 days after the last study drug administration:
5. Male subjects (including men who have had vasectomies) with a pregnant partner must agree to use a condom from the first dosing until at least 90 days after the last study drug administration.
6. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
7. Capable of consent.
8. Consent to perform genotyping for CYP2D6.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results
2. Positive urine drug screen or urine cotinine test at screening.
3. History of allergic reactions to GC4419, DM, or other related drugs.
4. Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first DM administration.
5. Poor CYP2D6 metabolizers as determined by genetic testing.
6. Positive pregnancy test at screening.
7. Any reason which, in the opinion of the Principal Investigator, would prevent the subject from participating in the study.
8. Clinically significant ECG abnormalities or vital sign abnormalities
9. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit
10. History of significant drug abuse
11. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
12. Use of medication other than hormonal contraceptives and topical products without significant systemic absorption:
13. Donation of plasma within 7 days prior to dosing.
14. Breast-feeding subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for dextromethorphan (DM) (in plasma): AUC0-t | Pre-dose on Day 1, and at 0.5, 1 (immediately prior to the end of GC4419 infusion), 2, 3, 4, 6, 8, 12, and 24 hours after the start of infusion
Pharmacokinetic (PK) profile for dextromethorphan (DM) (in plasma): AUC0-inf | Pre-dose on Day 1, and at 0.5, 1 (immediately prior to the end of GC4419 infusion), 2, 3, 4, 6, 8, 12, and 24 hours after the start of infusion
Pharmacokinetic (PK) profile for dextromethorphan (DM) (in plasma): Cmax | Pre-dose on Day 1, and at 0.5, 1 (immediately prior to the end of GC4419 infusion), 2, 3, 4, 6, 8, 12, and 24 hours after the start of infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Inventiv Health Clinical - Research Pharmacy Unit, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No